CLINICAL TRIAL: NCT06142812
Title: Gamification in the Classroom: Kahoot as a Tool for University Teaching Innovation.
Brief Title: Gamification in the University Classroom.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: -UJA
Record Dates: First submitted 2023-11-15; First posted 2023-11-22 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: University Student

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Students will be required to log in with a Pin number using a nickname that allows them to remain anonymous. Questions will be displayed on a large screen with four graphic shapes along with a countdown timer, and students will respond using their internet-enabled digital device. Students will choose, from four options, the possible answer by selecting the graphical shape, which they believe is correct, and will receive instant feedback accordingly. After each question, the game will rank players based on their speed and accuracy. The system will award a higher score to the student who enters the correct answer first. At the end of the quiz, the names of the top five players will be displayed on the leaderboard. The results can then be downloaded to highlight problematic questions and identify students who may be struggling.
  Interventions: Other: Kahoot!™ Group

INTERVENTIONS:
Other: Kahoot!™ Group — The theoretical concepts of each subject were taught over a period of four months, with a total duration of 30 hours. Of the total theoretical concepts of the subject, 50% were randomly selected to receive reinforcement through Kahoot! Each of the theoretical concepts chosen at random was consolidated through a Kahoot! questionnaire. which consisted of 15 questions, with three answer options. This questionnaire was administered at the end of the theoretical explanation of each section, with the objective of strengthening the learning of the contents just presented. After students answered each question in Kahoot!, the teacher clarified any questions related to that question and provided explanations as to why one answer was correct and the other two were incorrect. This process offered immediate feedback to students.

SUMMARY:
This article aims to demonstrate the results of a study on the implementation of Kahoot as a gamification tool in university education. The objectives of this article are: to promote teaching by integrating the use of Kahoot to motivate students and increase their degree of interest and know the students' abilities. opinions on the implementation of this Gamification tool to teach grammar. The study uses a quasi-experimental research design over a four-month period observing variables such as attention, concentration and creativity, as well as social and personal skills.

ELIGIBILITY:
Inclusion Criteria:

* University participants who were enrolled in the second year of the Physiotherapy Degree at the University of Jaén will be included.
* Study Period: Those participants who were available and participated in the study from September to December 2022 were considered.

Exclusion Criteria:

* University students who did not provide informed consent according to the study's ethical guidelines.
* Enrolled in at least one subject from another academic year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
D2 test | Up to twelve weeks
  Evaluates selective attention and concentration in the school context. The participant's task is to check carefully, starting from left to right, what is written on each line and must mark all the letters that have two small lines (two below, two above or one below and one above) with a "d". ". These elements are considered relevant. The other combinations (the "d" and the "p", with and without dashes) are considered irrelevant and should not be marked. The participant has 20 s for each line. This test has shown excellent reliability, with ranges between 0.90 and 0.97 for both Cronbach's α and the test-retest, and has also shown convergent and divergent validity.
Creative intelligence test (CREA) | Up to twelve weeks
  Evaluates creative intelligence by asking questions about an image. The participant, without opening the image, fills in spaces with provided data. Then the image is shown, and the task is to ask as many questions as possible. Questions are evaluated according to specific guidelines, scoring positively appropriate questions and penalizing decontextualized ones. Additional points are awarded for compound questions. The final score is calculated considering the number of questions, omissions, canceled answers and extra points. A high score (75-99 points) indicates excellent creative abilities, medium (26-74 points) indicates a moderate level of creativity, and low (1-25 points) suggests limited creative ability.
The ability subscale of the SEQ developed by Kember & Leung | Up to twelve weeks
  Will be used to collect data on students' reflections on the development of their generic abilities. It consists of 16 items that measure eight aspects of ability: critical thinking (2 items), creative thinking (2 items), self-managed learning (2 items), adaptability (2 items), problem solving (2 items), communication skills . (2 items), interpersonal skills and group work (2 items) and computer knowledge (2 items). Responses were recorded on a five-point Likert scale ranging from 5 ("strongly agree") to 1 ("strongly disagree"). The questionnaire also contains two open-ended questions to gather feedback on the best aspect and the one that needs improvement the most. In this study, the reliability of the ability subscale was high, with Cronbach's alphas of 0.86 and 0.92.

CONTACTS AND LOCATIONS:
Locations (1):
- Agustín Aibar Almazán, Jaén, Spain

IPD SHARING:
Plan to Share IPD: No